CLINICAL TRIAL: NCT03400605
Title: Parkdale Infant Nutrition Security Targeted Evaluation Project (PINSTEP): Formative Research (Objective 3-Infant Feeding)
Brief Title: Parkdale Infant Nutrition Security Targeted Evaluation Project: Infant Feeding
Acronym: PINSTEP-3
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Sellen, Professor, University of Toronto
Other Study IDs: 34482-3
Record Dates: First submitted 2017-12-08; First posted 2018-01-17 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Infant Nutrition; Vulnerable Population; Complementary Feeding; Food Security
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Program Clients: Parkdale Parents' Primary Prevention Project (5P's) clients
  Interventions: Other: Infant feeding questionnaire

INTERVENTIONS:
Other: Infant feeding questionnaire — Prospective infant feeding questionnaire administered over the telephone or in-person at 2 weeks and at 2, 4 and 6 months postpartum

SUMMARY:
In Toronto Ontario, the Parkdale Community Health Centre operates a community outreach program entitled Parkdale Parents' Primary Prevention Project (5P's). The 5P's provides weekly pre- and post-natal support and education programs for clients. This includes an infant feeding program for mothers with infants 0-6 months (Feeding Tiny Souls). The 5P's has a diverse client-base; the program is aimed at women who are in challenging life circumstances, therefore, clients may include low-income or single mothers and newcomers to Canada.

The aim of this project is to investigate the incidence, duration and exclusivity of breastfeeding and timely complementary feeding based on level of maternal participation in components of a pre and postnatal community outreach program. Exploring infant feeding practices is an evaluation component that will not only characterize infant feeding practices within a vulnerable population, but will elucidate whether there are areas of concern that need to be expanded upon within pre or postnatal programming. A prospective infant feeding questionnaire will be administered to participants at 2 weeks and at 2, 4 and 6 months postpartum. The study population will consist of women who enrolled in 5P's prenatally. The hypothesis is that exclusive breastfeeding rates will be low, but higher breastfeeding rates will be observed among women who utilize provided postnatal services more readily.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Parkdale Parents' Primary Prevention Project (5P's) prenatally
* Enrolled prenatally in 5P's as of August 17, 2017 onwards

Exclusion Criteria:

* Only enrolled in Parkdale Parents' Primary Prevention Project (5P's) postnatally
* Unavailable to participate in infant feeding questionnaire by telephone or in-person during 5P's programming

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Clients enrolled in Parkdale Parents' Primary Prevention Project (5P's) at Parkdale Community Health Centre in Toronto, Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding as assessed by responses to an infant feeding questionnaire | birth to 6 months postpartum
  Reported exclusive breastfeeding from birth to 6 months in response to a prospective infant feeding questionnaire

SECONDARY OUTCOMES:
Breastfeeding initiation as assessed by responses to an infant feeding questionnaire administered at 2 weeks postpartum | birth to 2 weeks postpartum
  Reported started breastfeeding at birth in response to a prospective infant feeding questionnaire
Breastfeeding duration as assessed by responses to an infant feeding questionnaire administered at 2 weeks and 2, 4 and 6 months postpartum | birth to 6 months
  Reported length of breastfeeding from birth to 6 months in response to a prospective infant feeding questionnaire
Introduction of complementary foods as assessed by responses to an infant feeding questionnaire administered at 2 weeks and 2, 4 and 6 months postpartum | birth to 6 months
  Reported timing of the introduction of complementary foods from birth to 6 months in response to a prospective infant feeding questionnaire
Types of complementary foods introduced as assessed by responses to a prospective infant feeding questionnaire administered at 2 weeks and 2, 4 and 6 months postpartum | birth to 6 months
  Reported types of foods introduced to infants from birth to 6 months in response to an infant feeding questionnaire
Vitamin and mineral supplementation as assessed by responses to an infant feeding questionnaire administered at 2 weeks and 2, 4 and 6 months postpartum | birth to 6 months
  Reported provision of vitamin or mineral supplementation to infants from birth to 6 months in response to a prospective infant feeding questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jane Francis, MSc, Principal Investigator — University of Toronto
Locations (1):
- Parkdale Community Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Francis J, Mildon A, Stewart S, Underhill B, Ismail S, Di Ruggiero E, Tarasuk V, Sellen DW, O'Connor DL. Breastfeeding rates are high in a prenatal community support program targeting vulnerable women and offering enhanced postnatal lactation support: a prospective cohort study. Int J Equity Health. 2021 Mar 3;20(1):71. doi: 10.1186/s12939-021-01386-6. PMID 33658034
- [Derived] Mildon A, Francis J, Stewart S, Underhill B, Ng YM, Rousseau C, Di Ruggiero E, Dennis CL, Kiss A, O'Connor DL, Sellen DW. Associations between use of expressed human milk at 2 weeks postpartum and human milk feeding practices to 6 months: a prospective cohort study with vulnerable women in Toronto, Canada. BMJ Open. 2022 Jun 8;12(6):e055830. doi: 10.1136/bmjopen-2021-055830. PMID 35676013
- See also: Related Info — https://equityhealthj.biomedcentral.com/articles/10.1186/s12939-021-01386-6